CLINICAL TRIAL: NCT02636075
Title: "Parathyroid Tissues Anatomic Localizations Are Displaced Downward in Parathyroid Hyperplasia Cases"
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Erhan Aysan, Head of the Department of General Surgery, SB Istanbul Education and Research Hospital
Other Study IDs: 123456ab
Record Dates: First submitted 2015-12-05; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Parathyroid Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Upper 1/3 of thyroid tissue
- Middle 1/3 of thyroid tissue
- Lower 1/3 of thyroid tissue
- Below thyroid tissue

SUMMARY:
This study investigates if Parathyroid Tissues Anatomic Localizations Are Displaced Downward in Parathyroid Hyperplasia Cases or not.

DETAILED DESCRIPTION:
Parathyroid tissues gets heavier when they become Hyperplasia. Because of this weight change, they change their normal anatomic positions. 125 patients who have been operated earlier will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone an operation due to parathyroid hyperplasia

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: no limitaion
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Size of the thyroid tissue | one year
  Longitudinal size (in mm) of each parathyroid tissue according to its anatomical location (upper, middle or lower 1/3 of the thyroid gland or below the thyroid)

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Aysan, MD, Study Director — Vakıf Gureba University